CLINICAL TRIAL: NCT02912624
Title: Combining Conventional With Advanced Hemodynamic Parameters for Predicting the Outcome of Critically Ill Patients: a Pilot for a Registry
Brief Title: Simple Intensive Care Studies I (SICS-I)
Acronym: SICS-I
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, I.C.C. van der Horst, Associate professor, University Medical Center Groningen
Other Study IDs: 201500144
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness; Acute Disease; Shock
Keywords: Physical Examination; Diagnostic Imaging; Ultrasonography; Hemodynamics; Patient Outcome Assessment; Mortality
MeSH Terms: conditions — Critical Illness; Acute Disease; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Circulatory shock is a condition of generalized inadequate blood flow through the body, leading to insufficient tissue perfusion and inadequate delivery of oxygen and other nutrients, to the extent that tissues are damaged. Four basic mechanisms of circulatory failure are distinguished, caused by a scale of underlying illnesses: distributive, hypovolemic, obstructive and cardiogenic shock. The last three types are characterized by a low cardiac output and hypovolemia. Distributive shock is characterized by peripheral circulation failure, with a low systemic vascular resistance, a disturbed microcirculation and a high cardiac output. Frequently, these forms overlap.

Shock is a common problem in the intensive care unit (ICU) as it affects about one third of the patients. Septic shock appears to be the most common type, followed by cardiogenic and hypovolemic shock. The diagnosis of shock is based on clinical examination with use of well-known circulatory parameters such as blood pressure and heart rate; biochemical parameters such as lactate and direct (semi-)invasive measurement of cardiac output and other variables.

Since cardiac output is an important determinant of oxygen delivery, many different methods of measuring cardiac output have been suggested. These methods range from non-invasive to invasive measurements with central lining. The most invasive method, the pulmonary artery catheter (PAC) has long been considered the optimal form of monitoring cardiac output by using thermodilution. However, this technique is associated with adverse events, such as bleeding, and there is no clear evidence of improved outcome. Therefore, numerous other techniques have been proposed, ranging from systems that use the dilution technique but only require central venous and peripheral artery lines; to less invasive tools that estimate cardiac output based on the arterial pressure waveform; and to non-invasive echocardiography.

Despite technical advances, much remains unknown about the value of conventionally used hemodynamic parameters for estimating cardiac output. A distinction between macro- and microcirculatory parameters can be made. Commonly used macro-circulatory parameters are heart rate, systolic and diastolic blood pressure, mean arterial pressure and central venous pressure. Lactate is used as a proxy for microcirculatory status. Over the years several other measurements have been suggested to improve insight in the hemodynamics of a certain patient or a group of patients. Skin temperature, capillary refill, mottling score and urinary output are used for hemodynamic assessment of the peripheral circulation and tissue perfusion. Most of these parameters have not been evaluated in a large prospective study and especially a combination of all these parameters has not directly been correlated to cardiac output.

More knowledge on the predictive value of all hemodynamic parameters in estimating cardiac output could assist physicians in earlier detection of impaired hemodynamics without the need for invasive or advanced methods. In this study the investigators aim to evaluate all hemodynamic parameters in a large unselected population of critically ill patients and to correlate them to cardiac output.

Purpose:

The purpose of this study is to create an infrastructure for a registry flexible to incorporate temporarily added specific research questions on the outcome of critically ill patients.

DETAILED DESCRIPTION:
Registry procedures:

Eligible patients will be included within 24 hours after their arrival on the Intensive Care Unit. After inclusion all study parameters will be obtained once through physical examination combined with transthoracic echocardiography. Mortality will be assessed at 90 days after admission. In addition, mortality follow-up will be cut-off at 7 and 30 days after admission.

Monitoring:

Monitoring will be performed by independent researchers of the department of anaesthesiology of the UMCG. Audits are planned to take place once a year.

Quality assurance plan:

Recruitment:

Inclusion of patients and measurements of variables (both conventional hemodynamic variables and cardiac output) will be performed by the study coordinator or a co-researcher under supervision and responsibility of the principle investigator. Informed consent will be obtained.

Source data verification:

At inclusion all conventional hemodynamic variables are derived by physical examination and recording data from the basic hemodynamic monitoring (Philips ImageVue monitor with tracing of heart rate, electrocardiogram (ECG), SpO2, arterial pressure from arterial line pressure measurement and/or from non-invasively blood pressure monitoring). In addition, a transthoracic echocardiography (TTE) will be performed to non-invasively determine the cardiac output by using the diameter of the aortic annulus, the velocity time integral (VTI) of the Doppler flow and the heart rate. All variables are predefined (see data dictionary) to standardize all measurements by student researchers.

For the performance of the TTE the student researchers will be trained to visualize the parasternal 2 chamber view, apical 4 and 5 chamber view according to the international standards (ACC/ESC) and to measure the left ventricular outflow tract VTI and the diameter of the aortic annulus. The training was given by an experienced cardiologist-intensivist. All measurements were validated by an echocardiography technician (core laboratory) who was blinded for all other measurement outcomes. General patient characteristics and laboratory measurements were recorded from electronic patient charts and the APACHE II and IV, Simplified Acute Physiology Score II (SAPS) scores are extracted from our local National Intensive Care Evaluation database. Follow-up of all-cause mortality is acquired using the municipal personal records database.

Standard Operation Procedures

Data collection:

Within 24 hours of ICU admission, all hemodynamic variables will be obtained through a onetime physical examination combined with transthoracic echocardiography. Other variables (i.e. lab values) will be obtained from the electronic patient charts at a later moment. The rationale and specific details of measuring each variable are described extensively below.

Systemic circulatory variables:

* Cardiac output (CO): it will be measured by transthoracic echocardiography, performed by different trained researchers. Both cardiac output and cardiac index (i.e. cardiac output corrected for body surface area) will be calculated.
* Stroke volume (SV): this will be automatically calculated by dividing cardiac output by heart rate, both measured by transthoracic echocardiography.
* Heart rate (HR): it will be recorded from the bedside electrocardiographic monitor. In case of an irregular rhythm (i.e. atrial fibrillation) the investigators will use the mean heart rate over a minute. Apart from heart rate the presence of atrial fibrillation will be recorded.
* Systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean arterial pressure (MAP): these will be obtained by intravascular measurement using an arterial line, which is part of usual care. To allow for comparison, these variables will also be measured using a sphygmomanometer. In the latter case, mean arterial pressure will be calculated using the following formula: MAP = (SBP + 2*DBP)/3
* Central venous pressure (CVP): this will be recorded in case a central venous line is present in the internal jugular or subclavian vene.

Micro- and peripheral circulatory variables:

* Capillary refill time (CRT): this will be measured after 15 seconds of exerting firm pressure preferably on the distal phalanx of the index finger and on the central part of the knee. The original upper limit of a normal CRT was considered to be 2 seconds by Champions' Trauma score. However Schriger and Baraff examined CRT in a healthy population and discovered it to be age and temperature dependent, with an upper limit for healthy older adults of 4.5 seconds. In a recent study Ait-Oufella et al found that an index CRT upper limit of 2.4 seconds is predictive of 14 day mortality in septic shock patients. The investigators will therefore both use a cut-off value of 4,5 seconds and a continuous measure of CRT.
* Skin temperature (Tskin): this will be measured subjectively and objectively. The subjective measure will be conducted by palpating the patient's extremities. A distinction between either 'warm' or 'cold' will be made using the dorsal surface of the hands of the examiner. Patients will be considered to have 'cold' skin extremities if all examined extremities are considered cool, or if only the lower extremities are cool despite warm upper extremities.

To objectify the skin temperature, the use of a central-to-peripheral and peripheral-to-ambient temperature difference (respectively dTc-p and dTp-a) or the forearm-to-finger skin-temperature gradient (Tskin-diff) have been proposed in literature. The investigators will make use of the central-to-peripheral measurements:

* Central-to-peripheral temperature difference (dTc-p): to measure this difference the investigators will compare bladder temperature, as measured by a bladder thermistor catheter, with foot temperature, measured by a skin probe (DeRoyal Skin Temperature Sensor product nr 81-010400EU) on either the left or the right big toe. The investigators will use bladder temperature as a surrogate for central temperature, and toe temperature as a peripheral measure. In literature a temperature difference of either 5°C or 7 °C is generally used as an upper limit. The investigators will therefore regard values higher than 7°C as abnormal.
* The mottling score: this score was described by Ait-Oufella et al in 2011. Mottling is the patchy discoloration of the skin caused by microcirculatory dysfunction. It usually involves the area around the knee. The Mottling score ranges from 0 -5, depending on the extensiveness of the mottled area. A score of 0-1 is regarded mild, 2-3 moderate and 4-5 severe.
* Urine output (ml/kg/h): this is also measured as part of regular care. The investigators will use both the urine output over the hour before examination and the mean urine output per hour, calculated using the six hours prior to the physical examination. If these data are unavailable, the mean urine output of the previous hour(s) will be calculated depending on the available data. In patients with pre-existing renal failure the urinary output will not be used.

Other variables:

* Respiratory rate: this will be recorded of the bedside electrocardiographic monitor. If a patient is on mechanical ventilation, see below.
* AVPU scale: this can be used to obtain a quick impression of a patients state of consciousness and consists of the options: 'Alert', 'responsive to Voice', 'responsive to Pain' and 'Unresponsive.' It is often applied in the emergency room and the general wards as part of the 'MEWS' (Modified Early Warning Score). The investigators will score the AVPU scale as a separate item.
* Cardiac murmurs: the investigators will auscultate the heart for the presence of a murmur. The potential cause of a cardiac murmur ranges from completely innocent to advanced valvular disease, each with its own distinctive characteristics. For study purposes, the investigators will score this item as: present or absent.
* Crepitations: the investigators will auscultate the lungs for crepitations, or crackles. In general a distinction between in- or expiratory and fine or coarse crepitations is made. Crepitations can be a symptom of several diseases, ranging from pneumonia and pulmonary edema to interstitial lung fibrosis. For study purposes, the investigators will only make a distinction in: present or absent.
* Serum lactate, creatinine and hemoglobin: these are determined as part of regular care. For study purposes the investigators will use the value closest to our examination. Other biochemical values will also be recorded.
* Mechanical ventilation: data on the presence and type of mechanical ventilation will be gathered, as well as basic information on respiratory conditions (i.e. PEEP and respiratory rate). Note: in case of mechanical ventilation the value 'respiratory rate' will be filled in twice in the CRF. If both values are the same, it will be assumed that the patient breathes at a machine-set respiratory rate. If they differ, spontaneous breathing will be assumed.
* Inotrope-, vasopressor and sedative use: any inotrope or vasopressin requirement, type, dose and speed will be recorded.
* Estimations of pump function and peripheral circulation: an estimation will be made, either by a member of the treating team, or by the researcher.

After the physical examination has been performed, information on the following general characteristics will be extracted from patient files: demographic data, diagnoses and severity of illness as evaluated by the APACHE II and IV scores, Simplified Acute Physiology Score II (SAPS) and the Sequential Organ Failure Assessment (SOFA). Furthermore the investigators will collect EMV scores, lab values (details are described above), urine output (details are described above), routine admission ECG's and routine admission thorax photo's. After 90 days the investigators will assess the patient files again to gather information on total ICU stay in days and 7-, 28- and 90-day mortality.

Data management:

Data will be recorded using OpenClinica and transferred for analysis. After transfer from OpenClinica, all data will be managed in a database created using Stata version 14.1 (StataCorp, College Station, TX) All study subjects will receive a study subject ID, compiled of the study name and their inclusion number. This study subject ID will be used in both OpenClinica and Stata. Only a researcher with 'study director' account properties in OpenClinica will be able to link study subject ID to patient number. Images will be saved anonymously and will be coded in a systematic fashion, using the study subject ID, session number, and image contents.

Sample size assessment:

There are no previous studies with data on including a combination of all available hemodynamic variables into one model estimating cardiac output and mortality. This makes it difficult to calculate sample size. The investigators will therefore make an estimation based on the number of ICU admissions per year. Each year 3000 patients are admitted to one of four ICU units. Approximately 1500 of these admissions are unplanned emergency admissions. The investigators estimate that half of these unplanned admissions fulfill the inclusion criteria. This leaves 750 patients eligible for inclusion. However, the investigators assume that they will not be able to include all eligible patients for logistic and practical reasons. Therefore the investigators aim to include 400 patients per year. With emergency admission critical care mortality approaching 25% this will enable us to include at least ten variables in the final model for predicting mortality (acknowledging that at least 10 events are necessary for each variable included in the final model). We will describe the power and detectable difference in a detailed statistical analysis plan (SAP).

Plan for missing data:

Primary analyses will be performed with imputation for missing data using multiple imputations. Robustness of conclusions will be checked by secondary sensitivity analyses only including available data. We will describe additional information in a detailed statistical analysis plan.

Statistical analysis plan:

The investigators will use the general characteristics to create a baseline table. Statistical analyses will be performed using the Stata (StataCorp, College Station, TX). Data will be presented as means with standard deviation if normally distributed or as medians with ranges in case of skewed data.

Univariate analyses will be conducted and all variables with p<0.1 will be included in the multivariate models. Multivariate analyses will be conducted using a stepwise model. Cardiac output will be modeled using linear regression and mortality will be modeled using logistic regression. All analyses will be adjusted for age and gender; other general characteristics will not be added to the model standardly. All analyses will be tested two-sided and p-values of less than 0.015 will be considered statistical significant. Multiplicity issues are described in our detailed SAP.

If sample size permits, the investigators will conduct an analysis in different subpopulations. Examples of subpopulations that may be eligible for further analysis are those with different types of shock (distributive, obstructive, hypovolemic, cardiogenic), CVVH, heart failure by any cause, myocardial infarction, atrial fibrillation or surgery versus no-surgery patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Emergency admission
* Expected stay > 24 hours

Exclusion Criteria:

* Age < 18 years
* Planned admission (either after surgery or for other reasons)
* Withdrawn or unable to obtain informed consent
* Continuous resuscitation efforts or mechanical circulatory support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in the adult Critical Care of the University of Groningen, University Medical Center Groningen, a tertiary teaching hospital in the Northern part of the Netherlands.
Sampling Method: Probability Sample
Enrollment: 1090 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2017-07-22 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
The association of a single or combination of clinical examination findings with cardiac index measured with transthoracic ultrasonography | Immediately
  Primary outcome of the basic study, answering our diagnostic research question
  We calculated cardiac index, which was derived from cardiac output. Cardiac output has been measured with the cardiac probe M3S of M4S with default cardiac imaging setting of the General Electric Vivid-S6 mobile ultrasound machine. Two views were obtained: the parasternal long axis (PLAX) and the apical five chamber view (AP5CH). The PLAX was used as the primary view to measure the left ventricular outflow tract (LVOT) diameter. The AP5CH view was used to measure the velocity time integral (VTI) using the pulse wave Doppler signal in the LVOT. Cardiac output was calculated on the ultrasound machine according to the formula: Cardiac output (L/min)=heart rate ∙VTI∙π∙(1/2∙LVOT)^2
  Clinical examination findings have been collected during a one-time physical examination, which is further specified at the study description section.
The association of all measured clinical examination findings, biochemical values and hemodynamic variables measured with transthoracic echocardiography with 90-day mortality | 90 days
  Primary outcome of the basic study, answering our prognostic research question.
  Clinical examination findings, as well are specified at the study description section.
  Biochemical values are serum lactate, creatinine and hemoglobine (see study description).
  Hemodynamic variables are obtained from advanced patient monitoring devices, such as invasive central venous or arterial blood pressures, echocardiographic measurements, etc.
  Follow-up on all-cause mortality will be obtained from the municipal personal records database. Analysis of mortality will be performed using time-to-event data (patients were censored at 90-days of follow-up).

SECONDARY OUTCOMES:
The diagnostic test accuracy of a single or a combination of clinical examination findings to diagnose a low, normal and high cardiac index measured with transthoracic echocardiography | Immediately
  Secondary outcome of the basic study, answering our diagnostic research question.
  For this outcome, we will determine the cut-offs as follows:
  1. Use a cardiac index cut-off of 2.2 L/min/m2
  2. Identify the optimal cut-off(s) for cardiac index. We will use dot plots to assess the distribution of cardiac index stratified by the presence or absence of each (combination of) clinical examination finding(s) that indicate hypoperfusion. We will conduct a logistic regression with the dichotomised clinical examination finding as dependent variable and cardiac index as independent variable, including the assumed covariate(s) of each finding, and compute receiver operating characteristic (ROC)-curves to identify the optimal cut-off(s).
The association and diagnostic test accuracy of a single or combination of clinical examination findings with cardiac index in clinically different patient subgroups | Immediately
  Secondary outcome of the basic study, answering our diagnostic research question.
  If the sample size permits, we will conduct subgroup analysis in different subpopulations. We will create the following subgroups in the basic study and test both our prognostic and diagnostic hypotheses on:
  * Subgroup 1: subdivide the population into three groups: no shock, shock associated with a low cardiac output, shock associated with a high cardiac output.
  * Subgroup 2: subdivide the population by underlying pathologies that could influence the haemodynamic measurements in a patient: Patients admitted due to cardiac arrest, myocardial infarction, after liver transplantation or liver failure, and severe sepsis. Patients admitted or known with heart failure, central nervous system pathologies, and severe chronic cardiovascular disease.
The association of clinical examination, biochemical and haemodynamic variables and 7- and 30-day mortality | 30 days
  Secondary outcome of the basic study, answering our prognostic research question.
  This will be a sensitivity analyses on different follow-up times of mortality.
The association of clinical examination, biochemical and haemodynamic variables that are not visible to caregivers with 90-day mortality | 90 days
  Secondary outcome of the basic study, answering our prognostic research question.
  Variables not visible to caregivers are some of our clinical examination findings and cardiac index measurements. Clinical examination findings that were not shared with caregivers, were: capillary refill times, mottling scores and peripheral temperature measurements.
The association of clinical examination, biochemical and haemodynamic variables with 90-day mortality in clinically different patient subgroups | 90 days
  Secondary outcome of the basic study, answering our prognostic research question.
  If the sample size permits, we will conduct subgroup analysis in different subpopulations. We will create the following subgroups in the basic study and test both our prognostic and diagnostic hypotheses on:
  * Subgroup 1: subdivide the population into three groups: no shock, shock associated with a low cardiac output, shock associated with a high cardiac output.
  * Subgroup 2: subdivide the population by underlying pathologies that could influence the haemodynamic measurements in a patient: Patients admitted due to cardiac arrest, myocardial infarction, after liver transplantation or liver failure, and severe sepsis. Patients admitted or known with heart failure, central nervous system pathologies, and severe chronic cardiovascular disease.

OTHER OUTCOMES:
The association between clinical, biochemical and haemodynamic variables and tissue (muscle) StO2 at the knee measured by near-infrared spectroscopy (NIRS) with the Inspectra StO2 tissue oxygenation monitor | Immediately
  Substudy 1 - primary outcome
  StO2 was measured by NIRS with the Inspectra StO2 tissue oxygenation monitor, model 650 (Hutchinson Technology, Inc., Hutchinson, Minnesota, USA). We used a 15-mm probe to measure the StO2 at a depth of 14mm at two sites: the thenar eminence and the distal end of the vastus medialis muscle. The average StO2 value was calculated over 30 seconds after one minute of signal stabilisation.
The association between clinical, biochemical and haemodynamic variables and tissue (muscle) StO2 at the thenar muscle measured by near-infrared spectroscopy (NIRS) with the Inspectra StO2 tissue oxygenation monitor | Immediately
  Substudy 1 - secondary outcome
The association between tissue (muscle) StO2 measured by NIRS and 90-day mortality | Immediately
  Substudy 1 - secondary outcome
The diagnostic test accuracy of a B-profile measured with pulmonary ultrasonography compared to pulmonary oedema diagnosed by chest radiography | Immediately
  Substudy 2 - primary outcome
  Pulmonary ultrasound was conducted with the cardiac probe M3S of M4S with default cardiac imaging and maximal frequency (3.6 MHz) setting of the General Electric Vivid-S6 mobile ultrasound machine. We measured the presence or absence of B-lines at the six locations specified in the BLUE-protocol. The presence of a B-profile was defined by three or more B lines observed in at least three of the six BLUE points, or in two of the four lower BLUE points.
  Pulmonary oedema was diagnosed by the radiologist who reviewed chest radiographs as part of daily care. The radiologist was blinded for the variables collected in our study.
The diagnostic test accuracy of pulmonary crackles assessed with auscultation compared to pulmonary oedema diagnosed by chest radiography | Immediately
  Substudy 2 - primary outcome
The statistically and clinically significant difference in CO between patients with and without a B-profile measured with pulmonary ultrasonography | Immediately
  Substudy 2 - secondary outcome
  The presence of a B-profile was defined by three or more B lines observed in at least three of the six BLUE points, or in two of the four lower BLUE points.
The association between PEEP increase and cardiac output measured with transthoracic echocardiography | Immediately
  Substudy 3 - primary outcome
  Cardiac output was measured using the same ultrasound machine, probes, views and formulas as described in the primary outcome of the basic study.
  During the PEEP-challenge, an additional 10 cm H2O of PEEP was temporarily applied when supervised by the treating ICU physician. The PEEP was elevated for a maximum duration of 5 minutes during which the changes in cardiac output, heart rate, blood pressures and central venous pressure were recorded.
The association between RV-function measured by TAPSE or RV s' with transthoracic echocardiography and 90-day mortality | 90 days
  Substudy 4 - primary outcome
  TAPSE and RV s' have been measured with the cardiac probe M3S of M4S with default cardiac imaging setting of the General Electric Vivid-S6 mobile ultrasound machine. Both measurements were obtained in the AP4CH view. TAPSE was assessed in M-mode, after placing the cursor on the junction of the tricuspid valve and the RV free wall. RV s' was assessed in the tissue velocity imaging mode highlighting the area of interest. The pulsed Doppler sample volume was placed at the tricuspid level of the RV free (i.e. lateral) wall and the longitudinal velocity of excursion was measured.
The association between RV-function measured by TAPSE or RV s' with transthoracic echocardiography and clinical examination findings and cardiac output measured with transthoracic echocardiography | Immediately
  Substudy 4 - secondary outcome
The association between peripheral blood flow measured at the common carotid, subclavian, and common femoral arteries and cardiac output, all measured with (transthoracic) echocardiography | Immediately
  Substudy 5 - primary outcome
  Common carotid artery, subclavian artery, and common femoral artery flows have been measured with the linear probe 8L or 9L and default carotid setting of the General Electric Vivid-S6 mobile ultrasound machine.
The association between a calculated proxy for abdominal organ blood flow and acute kidney injury (AKI) according to the KDIGO criteria or 90-day mortality | 90 days
  Substudy 5 - secondary outcome
  A proxy for abdominal flow was calculated by subtracting flow over both left and right carotid, subclavian and femoral arteries from the cardiac output.
  AKI was established and classified following the kidney disease: improving global outcomes (KDIGO) criteria. Urine output and serum creatinine measurements from the first 72 hours of inclusion were analysed to establish and classify AKI for each patient.
The level of agreement between cardiac output measured by the FloTrac and cardiac output measured with transthoracic echocardiography | 24 hours
  Substudy 6 - primary outcome
  Cardiac output has been estimated with the FloTrac (Edwards Lifesciences, Irvine, California, USA) and a monitor to compute stroke volume and cardiac output (Vigileo, Edwards Lifesciences, Irvine, California, USA). The FloTrac analyses the arterial pressure waveform to compute stroke volume and cardiac output. The estimated cardiac output was compared to the cardiac output measured with the General Electric Vivid-S6 mobile ultrasound machine.
The changes in levels of agreement when factors are present that might influence the FloTrac measurements of cardiac output | 24 hours
  Substudy 6 - secondary outcome
The association between changes in clinical examination findings over 24 hours and changes in cardiac output measured with transthoracic echocardiography | 24 hours
  Substudy 7 - primary outcome
  We repeated the measurements of the variables collected in the basic study, sub-study 2, and sub-study 4. We performed these measurements 24 hours (minimum 22 to maximum 26 hours) after the first measurement and calculated differences. The sign of the variable indicates whether a variable has either increased (positive number) or decreased (negative number).
The association between changes in clinical examination, biochemical, and hemodynamic variables over 24 hours and 90-day mortality | 90 days
  Substudy 7 - secondary outcome
The association between RV-volume overload measured by tricuspid insufficiency and RV-diameters measured with transthoracic echocardiography and AKI by the KDIGO criteria | Immediately
  Substudy 8 - primary outcome
  Right ventricle diameters and tricuspid regurgitation velocity have been measured with the cardiac probe M3S of M4S with default cardiac imaging setting of the General Electric Vivid-S6 mobile ultrasound machine. The measurements were obtained in the AP4CH view with a right ventricle centred view.
  AKI was established and classified following the kidney disease: improving global outcomes (KDIGO) criteria. Urine output and serum creatinine measurements from the first 72 hours of inclusion were analysed to establish and classify AKI for each patient.
The association between clinical, biochemical, and hemodynamic variables and the development of AKI according to the KDIGO criteria | Immediately
  Substudy 8 - primary outcome
The association between RV-volume overload measured by tricuspid insufficiency and RV diameters measured with transthoracic echocardiography and 90-day mortality | 90 days
  Substudy 8 - secondary outcome
The association between clinical, biochemical, and hemodynamic variables and the development of AKI regardless of the presence of pre-existent chronic kidney disease | Immediately
  Substudy 8 - secondary outcome
The diagnostic accuracy of fluid responsiveness assessed by changes in EtCO2, heart rate and blood pressure compared to the PLR test | Immediately
  Substudy 9 - primary outcome
  Every passive leg raising manoeuvre was conducted for a maximum duration of 60 seconds during which the changes in cardiac output, heart rate, blood pressures, central venous pressure, and EtCO2 were recorded. Fluid responsiveness was diagnosed when cardiac output increased with 15% after the PLR-test.
The diagnostic accuracy of fluid responsiveness assessed by a PLR test without lowering the head of the bed compared to the standard PLR test | Immediately
  Substudy 9 - primary outcome
  During the fluid responsiveness study, two different PLR tests were applied when supervised by the treating ICU physician.
The association between a temporary PEEP-increase and cardiac output measured with transthoracic echocardiography in fluid responders and fluid non-responders | Immediately
  Substudy 9 - secondary outcome
  Fluid responsiveness was diagnosed when cardiac output increased with 15% after the PLR-test. The PEEP-challenge was conducted in a similar manner as described in sub-study 3.
The diagnostic accuracy of a temporary PEEP-increase compared to the standard PLR test | Immediately
  Substudy 9 - secondary outcome
The diagnostic accuracy of a B-profile assessed with pulmonary ultrasonography compared to bilateral consolidations assessed on chest radiography for the diagnosis of ARDS | Immediately
  Substudy 10 - primary outcome
  ARDS will be defined according to the Berlin ARDS criteria: 1) presence of acute hypoxemic respiratory failure defined by a PaO2/FiO2 ratio < 300 mm Hg and PEEP ≥ 5 cm H2O; 2) onset within one week of clinical insult or worsening respiratory symptoms; 3) bilateral consolidations on chest radiography or CT-thorax.
The association between B-lines measured with pulmonary ultrasonography and clinical examination findings, biochemical values and hemodynamic variables | Immediately
  Substudy 10 - secondary outcome
  Clinical examination findings, as well are specified at the study description section.
  Biochemical values are serum lactate, creatinine and hemoglobine (see study description).
  Hemodynamic variables are obtained from advanced patient monitoring devices, such as invasive central venous or arterial blood pressures, echocardiographic measurements, etc.
The association between LV- and RV-myocardial strain measured by tissue Doppler imaging with transthoracic echocardiography and 90-day mortality | 90 days
  Substudy 11 - primary outcome
  Myocardial strain and myocardial strain rates have been measured with the cardiac probe M3S of M4S with default cardiac imaging setting of the General Electric Vivid-S6 mobile ultrasound machine. The measurements were obtained in the AP4CH window with a left ventricle and right ventricle centred view for left and right myocardial strain, respectively.
The association between LV- and RV-myocardial strain imaging and conventional CCUS measurements such as TAPSE, RV 's and cardiac output, all obtained with transthoracic echocardiography | Immediately
  Substudy 11 - secondary outcome
The level of agreement between myocardial strain measured by tissue Doppler imaging and myocardial strain rate measured by speckle tracking, both obtained with transthoracic echocardiography | Immediately
  Substudy 11 - secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Iwan CC van der Horst, M.D., Ph.D., Principal Investigator — University of Groningen, University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hiemstra B, Eck RJ, Koster G, Wetterslev J, Perner A, Pettila V, Snieder H, Hummel YM, Wiersema R, de Smet AMGA, Keus F, van der Horst ICC; SICS Study Group. Clinical examination, critical care ultrasonography and outcomes in the critically ill: cohort profile of the Simple Intensive Care Studies-I. BMJ Open. 2017 Sep 27;7(9):e017170. doi: 10.1136/bmjopen-2017-017170. PMID 28963297
- [Derived] Cox EGM, Wiersema R, Eck RJ, Kaufmann T, Granholm A, Vaara ST, Moller MH, van Bussel BCT, Snieder H, Pleijhuis RG, van der Horst ICC, Keus F. External Validation of Mortality Prediction Models for Critical Illness Reveals Preserved Discrimination but Poor Calibration. Crit Care Med. 2023 Jan 1;51(1):80-90. doi: 10.1097/CCM.0000000000005712. Epub 2022 Nov 15. PMID 36378565
- [Derived] Cox EGM, Koster G, Baron A, Kaufmann T, Eck RJ, Veenstra TC, Hiemstra B, Wong A, Kwee TC, Tulleken JE, Keus F, Wiersema R, van der Horst ICC; SICS Study Group. Should the ultrasound probe replace your stethoscope? A SICS-I sub-study comparing lung ultrasound and pulmonary auscultation in the critically ill. Crit Care. 2020 Jan 13;24(1):14. doi: 10.1186/s13054-019-2719-8. PMID 31931844
- [Derived] Koster G, Kaufmann T, Hiemstra B, Wiersema R, Vos ME, Dijkhuizen D, Wong A, Scheeren TWL, Hummel YM, Keus F, van der Horst ICC. Feasibility of cardiac output measurements in critically ill patients by medical students. Ultrasound J. 2020 Jan 8;12(1):1. doi: 10.1186/s13089-020-0152-5. PMID 31912438
- [Derived] Kaufmann T, Castela Forte J, Hiemstra B, Wiering MA, Grzegorczyk M, Epema AH, van der Horst ICC; SICS Study Group. A Bayesian Network Analysis of the Diagnostic Process and Its Accuracy to Determine How Clinicians Estimate Cardiac Function in Critically Ill Patients: Prospective Observational Cohort Study. JMIR Med Inform. 2019 Oct 30;7(4):e15358. doi: 10.2196/15358. PMID 31670697
- [Derived] Kaufmann T, Clement RP, Hiemstra B, Vos JJ, Scheeren TWL, Keus F, van der Horst ICC; SICS Study Group. Disagreement in cardiac output measurements between fourth-generation FloTrac and critical care ultrasonography in patients with circulatory shock: a prospective observational study. J Intensive Care. 2019 Apr 11;7:21. doi: 10.1186/s40560-019-0373-5. eCollection 2019. PMID 31011425

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT02912624/SAP_000.pdf